CLINICAL TRIAL: NCT03514940
Title: Perinatal Diagnosis of Fetal GIT Anomalies
Brief Title: Perinatal Diagnosis of GIT Anomalies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other); National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Assistant Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: GIT
Record Dates: First submitted 2018-04-22; First posted 2018-05-03 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Fetal Anomalies
MeSH Terms: conditions — Congenital Abnormalities | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound — second trimester us scan will be made to pregnant women

SUMMARY:
fetal gastro intestinal abnormalities can be accurately diagnosed in second trimester

DETAILED DESCRIPTION:
prenatal diagnosis of these anomalies allows for early postnatal interventions and implementation of treatment options

ELIGIBILITY:
Inclusion Criteria:

* pregnant women either primi or multigravida
* pregnant in 18- 24 weeks

Exclusion Criteria:

* first trimester pregnant ladies

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant females
Study Population: pregnant ladies either primi or multigravida
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2020-06-03 (Estimated); Study Completion 2020-07-07 (Estimated)

PRIMARY OUTCOMES:
The number of participants who will be diagnosed to have GIT anomalies | within 5 moths
  GIT anomalies that will be diagnosed by US and confirmed postnatal and managed operatively

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, M.s.c, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
results will be published